CLINICAL TRIAL: NCT00129675
Title: Development of a Imaging Marker for Parkinson's Disease Through Use of Dynamic SPECT Imaging With [123I] Beta-CIT in Individuals With Parkinson's Symptoms
Brief Title: Study of Individuals With Parkinson's Symptoms But in Whom There is Diagnostic Uncertainty
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institute for Neurodegenerative Disorders (Other)
Collaborators: Molecular NeuroImaging (Other)
Responsible Party: Principal Investigator, Danna Jennings, MD, Danna Jennings, MD, Institute for Neurodegenerative Disorders
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: Query-PD Study
Record Dates: First submitted 2005-08-11; First posted 2005-08-12 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Parkinsonian Syndrome
Keywords: parkinson; diagnosis
MeSH Terms: conditions — Parkinsonian Disorders; Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- [123I]ß CIT (Experimental): To assess [123I]ß CIT and SPECT imaging
  Interventions: Drug: [123I]ß CIT

INTERVENTIONS:
Drug: [123I]ß CIT — Single Photon Emission Computed Tomography
  SPECT imaging uses the single photon emissions from radioactive compounds that are (most commonly) injected into a patient and are metabolized by specific organs or body systems. SPECT imaging is performed by using a gamma camera to acquire multiple 2-D images (also called projections), from multiple angles. A computer is then used to apply a tomographic reconstruction algorithm to the multiple projections, yielding a 3-D dataset. This dataset may then be manipulated to show thin slices along any chosen axis of the body, similar to those obtained from other tomographic techniques, such as MRI, CT, and PET. The resulting SPECT images reflect body/organ function as opposed to specific anatomy of other imaging modalities such as CT or MRI.
  Other Names: SPECT imaging

SUMMARY:
The overall goal of this study is to evaluate the use of dopamine transporter (DAT) imaging as a diagnostic tool in subjects with early parkinsonian symptoms, in whom Parkinson's disease (PD) or parkinsonian syndrome (PS) is suspected, but the diagnosis remains unclear from a clinical standpoint.

DETAILED DESCRIPTION:
* Subjects will be referred to the Institute for Neurodegenerative Disorders (IND) by practicing general neurologists with genuine uncertainty regarding the subject's diagnosis.
* Subjects with suspected PD or PS will be evaluated clinically and with DAT imaging, using b-CIT and SPECT. The DAT imaging procedure will take place over two days:
* On the first day participants are injected with [123I]ß CIT, an investigational radioactive material that localizes in the brain. Study participants will also have a thorough neurologic examination and standard neuropsychological testing, including testing of memory, concentration, abstraction and visual spatial functions.
* Twenty-four hours later study participants return to the Institute for Neurodegenerative Disorders where an investigational scanning procedure will be used to obtain SPECT (single photon emission computed tomography) images of the brain.
* Subjects will be asked to return within 3 months following the imaging study to have a repeat neurological examination by the two study neurologists at IND.
* Subjects will be asked to return at about 6 months and possibly again at one year following the imaging study for a final clinical evaluation by one of the study neurologists at IND.

ELIGIBILITY:
Inclusion Criteria:

* Age >21
* Any parkinsonian or extrapyramidal symptoms
* Parkinsonian symptoms for < 2 years duration.
* No significant abnormalities on screening laboratory studies including: CBC, Chem-20 and urinalysis.
* Willingness to comply with study protocol.

Exclusion Criteria:

* Pregnancy
* Significant medical disease including abnormalities on screening biochemical or hematological labs or abnormal electrocardiogram (ECG).

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2003-02; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Comparison of the imaging diagnosis, based on visual analysis and quantitative analysis, to the clinical diagnosis of the investigator blinded to the imaging results | 5 years

SECONDARY OUTCOMES:
Comparison of the DAT imaging diagnosis, initial diagnosis by the movement disorder experts and referral neurologist diagnosis to the 'gold standard' diagnosis | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Danna L Jennings, MD, Principal Investigator — Institute for Neurodegenerative Disorders
Locations (1):
- Institute for Neurodegenerative Disorders, New Haven, Connecticut, United States